CLINICAL TRIAL: NCT00086593
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Study to Evaluate the Efficacy and Safety of a Flexible Dose of Lamotrigine Compared to Placebo as an Adjunctive Therapy to an Atypical Antipsychotic Agent(s) in Subjects With Schizophrenia
Brief Title: Study Of An FDA-approved Drug As Additional Therapy In Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101464
Record Dates: First submitted 2004-07-06; First posted 2004-07-08 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Schizophrenia
Keywords: adjunctive; atypical antipsychotics; add-on; Schizophrenia; psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Lamotrigine

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
This is a 12-week study for the treatment of chronic persistent symptoms in participants with schizophrenia. Participants on a stable, optimal dose of up to two atypical antipsychotics who fulfill the screening criteria will be randomized to receive either an FDA-approved drug or placebo in addition to the current treatment. Safety will be closely monitored through vital signs, various tests, and blood and urine samples.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with schizophrenia.
* Exhibits persistent positive symptoms that have persisted for a minimum of 3 months prior to screening.
* Continuously taking 1-2 specific atypical antipsychotics for a minimum of 3 months and must be on a stable dose for at least 1 month prior to entering the study.
* Participant or a legal guardian is able to understand and sign the consent form.

Exclusion criteria:

* PANSS (Positive and Negative Syndrome Score) total score increases or decreases by more than 20% between the Screening and Baseline visits.
* Predominant Axis I disorder other than schizophrenia within 6 months prior to screening.
* History of clinically significant or unstable medical disorder or treatment that would interfere with the study.
* History of autistic disorder or another pervasive developmental disorder, organic brain disease, dementia, stroke, epilepsy or a history of seizures requiring treatment (this does not include febrile seizures as a child), or those who have suffered a traumatic head injury.
* Taking psychotropic or primarily centrally active medication at screening.
* Use of antidepressant medications or mood stabilizers within 1 month of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2004-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total score of the Positive and Negative Symptom Scale (PANSS) at Week 12. | 12 Weeks

SECONDARY OUTCOMES:
- Efficacy - Change from baseline in PANSS positive symptoms at Week 12 - Change from baseline in the Scale for the Assessment of Negative Symptoms (SANS) at Week 12 - Change from baseline in PANSS general psychopathology symptoms at Week 12. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- United States (20):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Pico Rivera, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Niles, Illinois
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Madison, Wisconsin
- Canada (12):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Miramichi, New Brunswick
  - GSK Investigational Site, Dartmouth, Nova Scotia
  - GSK Investigational Site, Sydney, Nova Scotia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
- United Kingdom (5):
  - GSK Investigational Site, Bedford, Bedfordshire
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Hull

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 101464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register